CLINICAL TRIAL: NCT07353827
Title: A Prospective, Open-Label Clinical Study of FOLFOX-HAIC Combined With Donafenib and Pucotenlimab as First-Line Treatment for Unresectable Intrahepatic Cholangiocarcinoma
Brief Title: FOLFOX-HAIC Combined With Donafenib and Pucotenlimab as First-Line Treatment for Unresectable Intrahepatic Cholangiocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhongguo Zhou, Principal Investigator, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-688-01
Record Dates: First submitted 2026-01-04; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Intrahepatic Cholangiocarcinoma (Icc); Hepatic Arterial Infusion Chemotherapy
Keywords: Unresectable liver cancer; Hepatic arterial infusion chemotherapy; Oxaliplatin-based chemotherapy; Immune checkpoint inhibitor therapy; Targeted anti-angiogenic therapy; Phase II clinical trial
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension | interventions — donafenib; Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOLFOX-HAIC + Donafenib + Pucotenlimab (Experimental): Participants receive combination therapy in 21-day cycles:
  HAIC (FOLFOX): Hepatic Arterial Infusion Chemotherapy administered on Day 1 via a port-catheter system:
  Oxaliplatin: 85 mg/m^2 intra-arterial infusion (2 hours). Leucovorin: 400 mg/m^2 intra-arterial infusion (2 hours). Fluorouracil: 400 mg/m^2 bolus intra-arterial injection, followed by 2400 mg/m^2 continuous intra-arterial infusion over 46 hours.
  Pucotenlimab: 200 mg administered via intravenous (IV) infusion on Day 1. Donafenib: 0.2 g (200 mg) administered orally, twice daily (BID), continuously throughout the cycle.
  Treatment continues until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Procedure: hepatic arterial infusion chemotherapy (HAIC); Drug: Donafenib; Drug: Pucotenlimab; Drug: FOLFOX (5-fluorouracil, Leucovorin, Oxaliplatin)

INTERVENTIONS:
Procedure: hepatic arterial infusion chemotherapy (HAIC) — This intervention consists of a combination regimen including hepatic arterial infusion chemotherapy, targeted therapy, and immunotherapy for the treatment of unresectable intrahepatic cholangiocarcinoma. Hepatic arterial infusion chemotherapy is delivered through an implanted hepatic arterial catheter using a FOLFOX-based regimen, allowing high local drug concentrations within the liver while reducing systemic exposure. Donafenib, an oral multikinase inhibitor with anti-angiogenic activity, is administered continuously during treatment. Pucotenlimab, a programmed cell death protein-1 inhibitor, is administered by intravenous infusion to enhance antitumor immune responses. The combination is intended to achieve synergistic antitumor effects through regional cytotoxic chemotherapy, inhibition of tumor angiogenesis, and immune checkpoint blockade. Safety and antitumor activity of the regimen will be evaluated throughout the study period.
Drug: Donafenib — This intervention consists of a combination regimen including hepatic arterial infusion chemotherapy, targeted therapy, and immunotherapy for the treatment of unresectable intrahepatic cholangiocarcinoma. Hepatic arterial infusion chemotherapy is delivered through an implanted hepatic arterial catheter using a FOLFOX-based regimen, allowing high local drug concentrations within the liver while reducing systemic exposure. Donafenib, an oral multikinase inhibitor with anti-angiogenic activity, is administered continuously during treatment. Pucotenlimab, a programmed cell death protein-1 inhibitor, is administered by intravenous infusion to enhance antitumor immune responses. The combination is intended to achieve synergistic antitumor effects through regional cytotoxic chemotherapy, inhibition of tumor angiogenesis, and immune checkpoint blockade. Safety and antitumor activity of the regimen will be evaluated throughout the study period.
Drug: Pucotenlimab — This intervention consists of a combination regimen including hepatic arterial infusion chemotherapy, targeted therapy, and immunotherapy for the treatment of unresectable intrahepatic cholangiocarcinoma. Hepatic arterial infusion chemotherapy is delivered through an implanted hepatic arterial catheter using a FOLFOX-based regimen, allowing high local drug concentrations within the liver while reducing systemic exposure. Donafenib, an oral multikinase inhibitor with anti-angiogenic activity, is administered continuously during treatment. Pucotenlimab, a programmed cell death protein-1 inhibitor, is administered by intravenous infusion to enhance antitumor immune responses. The combination is intended to achieve synergistic antitumor effects through regional cytotoxic chemotherapy, inhibition of tumor angiogenesis, and immune checkpoint blockade. Safety and antitumor activity of the regimen will be evaluated throughout the study period.
Drug: FOLFOX (5-fluorouracil, Leucovorin, Oxaliplatin) — This intervention consists of a combination regimen including hepatic arterial infusion chemotherapy, targeted therapy, and immunotherapy for the treatment of unresectable intrahepatic cholangiocarcinoma. Hepatic arterial infusion chemotherapy is delivered through an implanted hepatic arterial catheter using a FOLFOX-based regimen, allowing high local drug concentrations within the liver while reducing systemic exposure. Donafenib, an oral multikinase inhibitor with anti-angiogenic activity, is administered continuously during treatment. Pucotenlimab, a programmed cell death protein-1 inhibitor, is administered by intravenous infusion to enhance antitumor immune responses. The combination is intended to achieve synergistic antitumor effects through regional cytotoxic chemotherapy, inhibition of tumor angiogenesis, and immune checkpoint blockade. Safety and antitumor activity of the regimen will be evaluated throughout the study period.

SUMMARY:
This is a prospective, open-label, single-arm phase II study designed to evaluate the efficacy and safety of FOLFOX-based hepatic arterial infusion chemotherapy (HAIC) in combination with donafenib and pucotenlimab as first-line treatment in patients with unresectable intrahepatic cholangiocarcinoma.

Eligible patients will receive FOLFOX-HAIC administered every three weeks together with oral donafenib and intravenous pucotenlimab. Tumor response will be assessed according to RECIST v1.1. The primary objective of the study is to determine the objective response rate, and secondary objectives include progression-free survival, overall survival, disease control rate, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 to 75 years.
* Histologically or clinically diagnosed Hepatocellular Carcinoma (HCC) according to AASLD or EASL guidelines.
* Disease stage classified as Barcelona Clinic Liver Cancer (BCLC) stage B (unresectable) or stage C.
* No prior systemic treatment for advanced HCC (treatment-naïve).
* At least one measurable lesion according to RECIST v1.1 criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Child-Pugh liver function class A (score 5-6).
* Life expectancy of at least 3 months.
* Adequate bone marrow function: Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, Platelets ≥ 75 × 10^9/L, and Hemoglobin ≥ 90 g/L.
* Adequate liver function: Total bilirubin ≤ 1.5 × ULN; ALT and AST ≤ 5 × ULN.
* Adequate renal function: Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min.
* Adequate coagulation function: INR ≤ 1.5 or PT ≤ 1.5 × ULN.
* Participants suitable for hepatic artery catheterization and HAIC treatment as assessed by the investigator.
* Willingness to provide written informed consent.

Exclusion Criteria:

* Known hypersensitivity or allergy to Oxaliplatin, Fluorouracil, Leucovorin, Donafenib, Pucotenlimab, or any of their excipients.
* Previous treatment with anti-PD-1/PD-L1 antibodies, anti-CTLA-4 antibodies, or other immunomodulatory agents.
* Diagnosis of other malignant tumors within the past 5 years (excluding cured basal cell carcinoma of the skin or carcinoma in situ of the cervix).
* Presence of central nervous system (CNS) metastases.
* Active, known, or suspected autoimmune disease (e.g., systemic lupus erythematosus, rheumatoid arthritis) requiring systemic treatment.
* History of gastrointestinal bleeding, esophageal or gastric varices with bleeding risk, or other active bleeding within 6 months prior to enrollment.
* Severe cardiovascular disease, including unstable angina, myocardial infarction within 6 months, or uncontrolled hypertension.
* Active infection requiring systemic antibiotic therapy.
* Hepatitis B virus (HBV) DNA > 2000 IU/mL (participants must receive antiviral treatment to suppress viral load).
* Known Human Immunodeficiency Virus (HIV) infection or active Syphilis infection.
* Anatomy unsuitable for hepatic arterial catheterization (e.g., severe vascular variation or occlusion).
* Pregnant or breastfeeding women.
* Any condition that, in the opinion of the investigator, would jeopardize the safety of the participant or the integrity of the study data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From baseline until disease progression or loss of clinical benefit, assessed approximately every 6 to 9 weeks, up to 2 years.
  The ORR is defined as the percentage of participants who achieve a confirmed Complete Response (CR) or Partial Response (PR). Efficacy will be evaluated by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From baseline up to approximately 2 years.
  Defined as the time from the first date of study treatment to the date of first documented disease progression per RECIST v1.1 or death from any cause, whichever occurs first.
Overall Survival (OS) | From baseline up to approximately 3 years.
  Defined as the time from the first date of study treatment to the date of death from any cause.
Disease Control Rate (DCR) | From baseline until disease progression, assessed approximately every 6 to 9 weeks, up to 2 years.
  Defined as the percentage of participants who achieve a confirmed Complete Response (CR), Partial Response (PR), or Stable Disease (SD) maintained for a specified minimum duration, according to RECIST v1.1.
Duration of Response (DoR) | From date of first response up to approximately 2 years.
  Defined as the time from the first documentation of objective response (CR or PR) to the first documentation of disease progression or death from any cause.
Safety (Adverse Events) | From the first dose of study treatment through 30 days after the last dose.
  Number of participants with treatment-related adverse events as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
Surgical Conversion Rate | From baseline up to approximately 2 years.
  The percentage of participants with initially unresectable disease who undergo successful surgical resection (R0 resection) following study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-san University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) will be made available upon request after publication of the study results.